CLINICAL TRIAL: NCT04274634
Title: The Oscillation of Crystalline and Intraocular Lenses: a Feasibility Study of the Lens' Movements in the Eye
Brief Title: The Oscillation of Crystalline and Intraocular Lenses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anglia Ruskin University (Other)
Collaborators: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OSCCIL
Record Dates: First submitted 2020-02-03; First posted 2020-02-18 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Marfan's Syndrome With Ocular Manifestations; Pseudoexfoliation Syndrome; Cataract; Phakodonesis; Ectopia Lentis
MeSH Terms: conditions — Exfoliation Syndrome; Cataract; Ectopia Lentis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Conditions with predisposition to lens oscillations: Marfan Syndrome and Pseudoexfoliation
- Age-matched with normal axial lengths
- Age-matched with extreme axial lengths
- Intraocular lens
- Pre- and post- cataract surgery
- Normals

SUMMARY:
The crystalline lens of the human eye helps to sharpen vision. There can be issues with the support/stability of the lens. This could be seen with the naked eye of an external observer or with the use of a slit lamp.

Certain eye conditions can predispose to issues with lens stability. If patients have stability issues with their natural lens- this would be termed as "phakodonesis". However, in patients who have had prior cataract surgery with implantation of an artificial lens (IOL)- this would be termed as "pseudophakodonesis". Eye conditions such as pseudoexfoliation or Marfan-syndrome can lead to unstable lens support- this can be detected if there are advanced stability issues.

However, small instability in the eye's would not be detected with present descriptive methods. The authors have designed a high-speed camera which is able to detect stability of the lens, especially during eye movements. The high-speed camera can detect variation in the change of light reflex from the lens and calculate the amount of lens instability/oscillation. The results (in normal eyes) of this high-speed camera has already been published in a peer-review journal. It is non-contact and measures lens movement. The test lasts less than 5 minutes.

Further research is required to assess the amount of lens oscillation (wobbling) in different eye populations - patients with previous cataract surgery (an artificial implant is used to replace the lens) or eye conditions (such as pseudoexfoliation, Marfan syndrome). The amount of lens stability has a role in the planning of further intraocular surgery - especially cataract extraction - however, at present, there is no approved quantitative measurement for this.

Participants will be recruited through Anglia Ruskin University (educational establishment), local community groups, and through Southend University Hospital eye clinics (NHS organisation). Participants' data will remain anonymous.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Able to read and understand the English language

Exclusion Criteria:

* Significant corneal scarring
* Taking medications that cause miosis (pupil constriction)
* Patients with no light perception
* Patients unable to open their eyes e.g. due to significant ptosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care, community sample
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of implementing a larger study | 1 year
  Criteria: number of eligible participants.This can then inform the sample size calculation for the larger study.

SECONDARY OUTCOMES:
Assessing lens oscillation amplitude in different patient populations using a non-invasive, high-speed camera | 1 year
  The measurement tool is a non-invasive, high-speed camera device that is used to assess lens oscillations has been made for this purpose by one of the co investigators. The device measures lens oscillations in a quantitative way, being much simpler and more accurate compared to previous qualitative assessments. The outcome measure, lens oscillation, is measured by: amplitude, which will be compared across the six patient population groups.
Assessing lens oscillation ("wobbliness") by oscillation frequency in different patient populations using a non-invasive, high-speed camera | 1 year
  The measurement tool is a non-invasive, high-speed camera device that is used to assess lens oscillations has been made for this purpose by one of the co investigators. The device measures lens oscillations in a quantitative way, being much simpler and more accurate compared to previous qualitative assessments. The outcome measure, lens oscillation, is measured by: oscillation frequency, which will be compared across the six patient population groups.
Assessing lens oscillation by damping ratio in different patient populations using a non-invasive, high-speed camera | 1 year
  The measurement tool is a non-invasive, high-speed camera device that is used to assess lens oscillations has been made for this purpose by one of the co investigators. The device measures lens oscillations in a quantitative way, being much simpler and more accurate compared to previous qualitative assessments. The outcome measure, lens oscillation, is measured by: damping ratio, which will be compared across the six patient population groups.
Assessing lens oscillation by the stationary time in different patient populations using a non-invasive, high-speed camera | 1 year
  The measurement tool is a non-invasive, high-speed camera device that is used to assess lens oscillations has been made for this purpose by one of the co investigators. The device measures lens oscillations in a quantitative way, being much simpler and more accurate compared to previous qualitative assessments. The outcome measure, lens oscillation, is measured by: stationary time, which will be compared across the six patient population groups.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Southend University Hospital NHS Foundation Trust, Southend-on-Sea, Essex
  - Vision and Eye Research Institute (VERI), Cambridge

IPD SHARING:
Plan to Share IPD: Undecided